CLINICAL TRIAL: NCT07004114
Title: The Effects of Neurocognitive Training on Pain, Proprioception, Injury Anxiety, and Functional and Neurocognitive Performance in Athletes With Chronic Ankle Instability
Brief Title: Effects of Neurocognitive Training on Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Ebru Tekin, Lecturer, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/13
Record Dates: First submitted 2025-05-17; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Chronic Ankle Instability; Balance; Neurocognitive
Keywords: Cognitive Load; Ankle Instability; RBT

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurocognitive training group (Experimental): Neurocognitive training is a program developed by incorporating motor learning strategies and cognitive challenges into neuromuscular training. Cognitive challenges included tasks requiring quick reactions, motor-motor or cognitive-motor tasks (dual-task), congruent and incongruent tasks, exercises combined with mathematical calculations (working memory), and response inhibition tasks.
  Interventions: Other: Neurocognitive training group
- Control group (No Intervention): The control group continued their training and no additional intervention was applied. Four weeks after their initial assessment, the same assessments were applied again with the study group.

INTERVENTIONS:
Other: Neurocognitive training group — Neurocognitive training is a rehabilitation approach that, unlike traditional treatment methods which primarily focus on improving physical performance, emphasizes cognitive functions and psychometric skills. It is a program developed by integrating motor learning strategies and cognitive challenges into neuromuscular training. These cognitive challenges include tasks requiring quick reactions, motor-motor or cognitive-motor tasks (dual-task), congruent and incongruent tasks, exercises involving mathematical calculations (working memory), and response inhibition tasks.
  Arms: Neurocognitive training group

SUMMARY:
Aim: This study aimed to investigate the effects of neurocognitive training on pain, proprioception, injury-related fear, functional, and neurocognitive performance in athletes with chronic ankle instability (CAI).

Materials and Methods: A total of 30 athletes with CAI, with a mean age of 11.10±1.06 years and residing in Balıkesir, were included in the study. Participants were randomly assigned into two groups using simple randomization: the intervention group (n=15) and the control group (n=15). Two participants from the control group were excluded from the final analyses due to missing post-intervention assessments. The intervention group received a neurocognitive training program conducted twice a week for four weeks, following an initial familiarization week. The training was progressively administered on flat ground, balance mat, BOSU, and inverted BOSU. Both groups were evaluated before and after the 4-week intervention using the following measures: the Identification of Functional Ankle Instability (IdFAI), the Cumberland Ankle Instability Tool (CAIT), pain intensity, proprioception, fear of re-injury, Y Balance Test (YBT), Side Hop Test, Reactive Balance Test (RBT), and Upper Extremity Choice Reaction Time Test.

Results: The results were analyzed.

ELIGIBILITY:
Inclusion Criteria:

Aged between 10 and 18 years

At least 2 years of active athletic participation

History of ankle sprain with at least 2 inflammatory symptoms (e.g., pain, swelling)

The most recent sprain occurred at least 3 months prior to the study start date

A score of 11 or above on the FABIT (Simon et al., 2012)

A score of ≤27 on the CAIT (Yin et al., 2022)

Willingness to participate in the study

Exclusion Criteria:

History of hip/pelvis, knee, or ankle surgery within the past year

History of ankle fracture

Diagnosis of a neurological disorder

Presence of vestibular disorders

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Functional Ankle Instability Assessment Using the Identification of Functional Ankle Instability Questionnaire (IDFAI) | from the beginning of the study until the end of the 4th week
  The IDFAI is a self-reported questionnaire consisting of 9 items designed to identify the presence and severity of functional ankle instability. Scores range from 0 to 37, with higher scores indicating greater instability. A score above 11 suggests the presence of instability. Scores are unitless numeric values representing the severity of symptoms and frequency of ankle sprains.
Functional Ankle Instability Evaluation Using the Cumberland Ankle Instability Tool (CAIT) | from the beginning of the study until the end of the 4th week
  The CAIT is a self-assessment tool with 9 items measuring subjective ankle instability. Scores range from 0 (severe instability) to 30 (no instability). A score of 27 or below indicates functional ankle instability. The score is a unitless numeric value that reflects the level of perceived instability and risk of recurrent sprains.
Pain Severity Assessment-Visual Analog Scale (VAS) | from the beginning of the study until the end of the 4th week
  The Visual Analog Scale (VAS) is a 10 cm line ranging from "No pain" to "Worst imaginable pain." Participants mark their pain intensity on the line, which is measured in centimeters to quantify pain severity. This unitless numeric score reflects pain intensity at rest, during training, and post-training in ankles with instability history.

OTHER OUTCOMES:
Proprioception Assessment with Reposition Test (Ankle Dorsiflexion and Plantarflexion Angles) | from the beginning of the study until the end of the 4th week
  Joint Position Sense test evaluates proprioception by measuring the accuracy of reproducing a passively positioned joint angle. The ankle dorsiflexion is set at 10°, and plantarflexion at 20°. The difference between target and reproduced angles is measured in degrees using a goniometer. Lower angular deviation indicates better proprioceptive accuracy.
The Sport Injury Anxiety Scale (SIAS) | from the beginning of the study until the end of the 4th week
  The Sport Injury Anxiety Scale (SIAS) was developed to assess the level of anxiety athletes experience after injury. The Turkish adaptation, validity, and reliability study of the scale was conducted by Caz et al. (2019) with university students participating in amateur sports. An increase in the average score obtained from the scale indicates a higher level of injury-related anxiety (Caz et al., 2019).
Postural Stability Measurement Using Multireha Portable Balance Device (Sway in Millimeters During Single-Leg Stance) | from the beginning of the study until the end of the 4th week
  Using the Multireha portable balance device, postural stability is assessed by measuring the average sway in millimeters in anterior, posterior, medial, and lateral directions during a single-leg stance on the unstable ankle side. Two trials of 30 seconds are conducted. Lower sway values indicate better postural stability.
Dynamic Balance Evaluation Using the Y Balance Test (YBT) | from the beginning of the study until the end of the 4th week
  YBT measures dynamic balance in three directions: anterior, posteromedial, and posterolateral. The composite score is calculated as (sum of three reach distances) / (3 x limb length) × 100, yielding a percentage. Higher percentages reflect better dynamic balance and postural control.
Functional Performance Assessment with the Lateral Hop Test | from the beginning of the study until the end of the 4th week
  Participants perform 10 lateral hops over a 30 cm distance on the affected limb as fast as possible. The shortest completion time of two trials, measured in seconds, is recorded. Lower times indicate better functional performance and ankle stability.
Reactive Balance Performance Using the Reactive Balance Test (RBT) with LED Light System | from the beginning of the study until the end of the 4th week
  RBT combines YBT setup with a smartphone-connected LED system. Participants respond to randomly illuminated lights by touching them quickly without losing balance. Performance metrics include visual-motor reaction time (milliseconds) and accuracy percentage. Two trials are conducted; the second trial is recorded for analysis. Lower reaction times and higher accuracy indicate better reactive balance.
Upper Extremity Choice Reaction Time Test | from the beginning of the study until the end of the 4th week
  Participants sit with dominant hand ready to press LED lights arranged on a table. Lights illuminate randomly every 0.5-2.5 seconds. Reaction time (milliseconds) and accuracy (number of correct responses) over one minute are recorded. This test evaluates selective attention and cognitive-motor processing speed.

CONTACTS AND LOCATIONS:
Locations (1):
- Balikesir University, Balıkesir, Bigadiç, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohammadi F. Comparison of 3 preventive methods to reduce the recurrence of ankle inversion sprains in male soccer players. Am J Sports Med. 2007 Jun;35(6):922-6. doi: 10.1177/0363546507299259. Epub 2007 Mar 22. PMID 17379918
- [Background] Walker JM, Brunst CL, Chaput M, Wohl TR, Grooms DR. Integrating neurocognitive challenges into injury prevention training: A clinical commentary. Phys Ther Sport. 2021 Sep;51:8-16. doi: 10.1016/j.ptsp.2021.05.005. Epub 2021 May 19. PMID 34153635
- [Background] 18) Tekin E, Ünver F. Klinik Nörobilişsel Fonksiyonel Performans Testleri: Geleneksel Derleme. Turkiye Klinikleri Journal of Sports Sciences, 2023;15(2).
- [Background] Tassignon B, Verschueren J, Delahunt E, Smith M, Vicenzino B, Verhagen E, Meeusen R. Criteria-Based Return to Sport Decision-Making Following Lateral Ankle Sprain Injury: a Systematic Review and Narrative Synthesis. Sports Med. 2019 Apr;49(4):601-619. doi: 10.1007/s40279-019-01071-3. PMID 30747379
- [Background] Verschueren J, Tassignon B, Verhagen E, Meeusen R. The interaction of acute physical fatigue with three traditional functional performance tests and the reactive balance test. Phys Ther Sport. 2021 May;49:188-195. doi: 10.1016/j.ptsp.2021.03.004. Epub 2021 Mar 17. PMID 33756239
- [Background] Simon J, Donahue M, Docherty C. Development of the Identification of Functional Ankle Instability (IdFAI). Foot Ankle Int. 2012 Sep;33(9):755-63. doi: 10.3113/FAI.2012.0755. PMID 22995264
- [Background] Plisky PJ, Gorman PP, Butler RJ, Kiesel KB, Underwood FB, Elkins B. The reliability of an instrumented device for measuring components of the star excursion balance test. N Am J Sports Phys Ther. 2009 May;4(2):92-9. PMID 21509114
- [Background] 13) Olsson L, Lund H, Henriksen M, Rogind H, Bliddal H, Danneskiold Samsøe B. Test-retest reliability of a knee joint position sense measurement method in sitting and prone position. Advances in Physiotherapy. 2004;6(1):37-47.
- [Background] Obuz T, Topcu ZG. The effects of exercises with a Pilates ball on balance, reaction time and dual-task performance of kindergarten children. J Comp Eff Res. 2022 Jun;11(8):583-593. doi: 10.2217/cer-2021-0293. Epub 2022 May 6. PMID 35514277
- [Background] Loizidis T, Nikodelis T, Bakas E, Kollias I. The effects of dry needling on pain relief and functional balance in patients with sub-chronic low back pain. J Back Musculoskelet Rehabil. 2020;33(6):953-959. doi: 10.3233/BMR-181265. PMID 32310156
- [Background] Hiller CE, Refshauge KM, Bundy AC, Herbert RD, Kilbreath SL. The Cumberland ankle instability tool: a report of validity and reliability testing. Arch Phys Med Rehabil. 2006 Sep;87(9):1235-41. doi: 10.1016/j.apmr.2006.05.022. PMID 16935061
- [Background] Hertel J. Functional instability following lateral ankle sprain. Sports Med. 2000 May;29(5):361-71. doi: 10.2165/00007256-200029050-00005. PMID 10840868
- [Background] Gribble PA, Delahunt E, Bleakley C, Caulfield B, Docherty C, Fourchet F, Fong DT, Hertel J, Hiller C, Kaminski T, McKeon P, Refshauge K, van der Wees P, Vicenzino B, Wikstrom E. Selection criteria for patients with chronic ankle instability in controlled research: a position statement of the International Ankle Consortium. Br J Sports Med. 2014 Jul;48(13):1014-8. doi: 10.1136/bjsports-2013-093175. Epub 2013 Nov 19. PMID 24255768
- [Background] Fong DT, Hong Y, Chan LK, Yung PS, Chan KM. A systematic review on ankle injury and ankle sprain in sports. Sports Med. 2007;37(1):73-94. doi: 10.2165/00007256-200737010-00006. PMID 17190537
- [Background] Engeroff T, Giesche F, Niederer D, Gerten S, Wilke J, Vogt L, Banzer W. Explaining Upper or Lower Extremity Crossover Effects of Visuomotor Choice Reaction Time Training. Percept Mot Skills. 2019 Aug;126(4):675-693. doi: 10.1177/0031512519841755. Epub 2019 Apr 30. PMID 31039674
- [Background] 4) Caz Ç, Kayhan RF, Bardakçı S. Spor Yaralanması Kaygı Ölçeği'nin Türkçeye Uyarlanması: Geçerlik ve Güvenirlik Çalışması. Spor Hekimliği Dergisi. 2019;54(1): 52-63
- [Background] Caldemeyer LE, Brown SM, Mulcahey MK. Neuromuscular training for the prevention of ankle sprains in female athletes: a systematic review. Phys Sportsmed. 2020 Nov;48(4):363-369. doi: 10.1080/00913847.2020.1732246. Epub 2020 Feb 28. PMID 32067546
- [Background] Cain MS, Ban RJ, Chen YP, Geil MD, Goerger BM, Linens SW. Four-Week Ankle-Rehabilitation Programs in Adolescent Athletes With Chronic Ankle Instability. J Athl Train. 2020 Aug 1;55(8):801-810. doi: 10.4085/1062-6050-41-19. PMID 32577737
- [Background] 1) Akca NK, Aydın G, Gümüş K. Lomber disk hernili hastaların vücut mekanikleri bilgi düzeyleri ile ağrı şiddeti arasındaki ilişki. Gümüşhane Üniversitesi Sağlık Bilimleri Dergisi. 2013;2(1):66-77.